CLINICAL TRIAL: NCT00198068
Title: Predictors of Pregnancy Outcome in Systemic Lupus Erythematosus (SLE) and Antiphospholipid Syndrome (APS)
Acronym: PROMISSE
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2014-309; R01AR049772 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus; Antiphospholipid Syndrome
Keywords: Pregnancy outcomes; Systemic lupus erythematosus; Antiphospholipid syndrome
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, whole blood, RNA, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: aPL+/SLE-: Positive antiphospholipid antibodies (aPL) defined as positive LAC and/or anti cardiolipin IgG/IgM >= 40 units and/or anti-beta 2 glycoprotein I IgG or IgM >= 40 units; no SLE
- Group 2: aPL+/SLE+: Positive antiphospholipid antibodies (aPL) defined as positive LAC and/or anti cardiolipin IgG/IgM >= 40 units and/or anti-beta 2 glycoprotein I IgG or IgM >= 40 units AND SLE defined as four or more American College of Rheumatology criteria for SLE.
- Group 3: aPL-/SLE+: No antiphospholipid antibodies; SLE defined as four or more American College of Rheumatology criteria for SLE.
- Group 4: aPL-/SLE-: Healthy controls: no antiphospholipid antibodies; no SLE

SUMMARY:
The PROMISSE Study is an observational study of 700 pregnant patients, enrolled at nine major clinical centers. The purpose of the study is 1) to determine whether certain proteins (called complement split products) that can injure healthy organs can be used to predict poor pregnancy outcome in patients with systemic lupus erythematosus (SLE) and anti-phospholipid syndrome (APS), and/or 2) to determine whether elevated levels of circulating antiangiogenic factors predict pregnancy complications in patients with aPL antibodies and/or SLE.

DETAILED DESCRIPTION:
Thrombosis and pregnancy loss are common features of systemic lupus erythematosus (SLE), particularly in the presence of antiphospholipid (aPL) antibodies. The in vivo mechanisms by which aPL antibodies lead to vascular events and, specifically, to recurrent fetal loss are largely unknown. Studies in a mouse model of antiphospholipid antibody syndrome (APS) indicate that in vivo complement activation is necessary for fetal loss caused by aPL antibodies. This study represents an effort to translate these research observations on the potential role of complement activation in the pathogenesis of aPL antibody-mediated pregnancy loss to a clinically relevant human study.

In addition, studies in humans and mice have shown 1) that the balance of circulating angiogenic and antiangiogenic factors predicts preeclampsia and fetal growth restriction in healthy women, 2) circulating antiangiogenic factors cause endothelial dysfunction and abnormal placental development in animal models, and 3) complement activation leads to elevated levels of circulating antiangiogenic factors and complement inhibition prevents increased levels of antiangiogenic factors, placental dysfunction and fetal growth restriction in a mouse model of APS. This study will permit testing the hypothesis that, like in healthy women, the balance of circulating angiogenic and antiangiogenic factors predict complications in women with SLE and APS and to translate the findings in animal models into humans.

The PROMISSE Study is a prospective observational study that will follow 700 pregnant patients who will be grouped and analyzed according to the presence or absence of aPL antibodies and preexisting SLE. The patients are followed regularly during the course of the pregnancy, collecting medical and obstetrical information as well as serial blood specimens for complement and cytokine assays. The data obtained will be analyzed and used to identify mechanisms and predictors of poor fetal outcome. We expect that the insights provided through this study will suggest means to prevent, arrest or modify these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient pregnant with live intrauterine pregnancy, as defined by positive test for elevated β-HCG, but ≤ 12 weeks by gestation (for subjects without aPL antibodies) and ≤18 weeks (for subjects with aPL antibodies)
* Patient between the ages of 18-45 and able to give informed consent, or age < 18 years with parental consent
* Hematocrit > 26%
* For APL positive:

  * aCL: IgG >= 40 GPL units; IgM >= 40 MPL units
  * Positive LAC (RVVT, Kaolin, dilute TTI or PTT LA)
  * Anti-β2GPI: IgG >= 40 GPL units; IgM >= 40 MPL units
* For control subjects:

  * At least one successful pregnancy
  * No history of fetal death (death of conceptus ≥ 10 weeks' gestation)
  * No more than 1 miscarriage < 10 weeks' gestation
  * No history of positive aPL in local lab or positive aPL in core labs at screening
  * Not currently a smoker
  * No medical problems requiring chronic treatment

Exclusion Criteria:

* Diabetes mellitus (Type I and Type II) antedating pregnancy
* Known or suspected hereditary complement deficiency (defined by CH50 = 0)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients identified by investigators at each study site
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2003-09; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Otherwise unexplained fetal death occurring after 12 weeks gestation | End of pregnancy
  Fetal death occurring after 12 weeks' gestation and not explained by chromosomal abnormalities, anatomic malformations, or congenital infections.
Neonatal death | Time of neonatal death
  Neonatal death prior to hospital discharge and due to complications of prematurity
Preterm delivery prior to 36 weeks' gestation | End of pregnancy
  Indicated preterm delivery prior to 36 weeks' gestation because of gestational hypertension, preeclampsia-eclampsia or placental insufficiency
Small for gestational age (SGA) <5th %ile | End of pregnancy
  Small for gestational age (SGA) <5th %ile in the absence of anatomical or chromosomal abnormalities and/or delivery before 36 weeks because of intrauterine growth restriction (IUGR).

SECONDARY OUTCOMES:
Gestational age | End of pregnancy
  Gestational age (weeks and days) at the end of pregnancy
Birth weight | End of pregnancy
  Birth weight
Number of days neonate requires positive pressure ventilation | Neonate discharge from hospital
  Number of days neonate requires positive pressure ventilation
Total number of days neonate is hospitalized | Neonate discharge from hospital
  Total number of days neonate is hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Jane E. Salmon, M.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (10):
- United States (8):
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - NYU Langone Medical Center/Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - University of Utah Salt Lake City, Salt Lake City, Utah
- Mt. Sinai Hospital, Toronto, Ontario, Canada
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Because the investigative team is still analyzing the data for biomarkers and genetics, the authors are not willing to make the data public at this time. Published study results can be found under Publications on the ClinicalTrials.gov site for this study.

REFERENCES:
- [Background] Girardi G, Redecha P, Salmon JE. Heparin prevents antiphospholipid antibody-induced fetal loss by inhibiting complement activation. Nat Med. 2004 Nov;10(11):1222-6. doi: 10.1038/nm1121. Epub 2004 Oct 17. PMID 15489858
- [Background] Girardi G, Berman J, Redecha P, Spruce L, Thurman JM, Kraus D, Hollmann TJ, Casali P, Caroll MC, Wetsel RA, Lambris JD, Holers VM, Salmon JE. Complement C5a receptors and neutrophils mediate fetal injury in the antiphospholipid syndrome. J Clin Invest. 2003 Dec;112(11):1644-54. doi: 10.1172/JCI18817. PMID 14660741
- [Background] Holers VM, Girardi G, Mo L, Guthridge JM, Molina H, Pierangeli SS, Espinola R, Xiaowei LE, Mao D, Vialpando CG, Salmon JE. Complement C3 activation is required for antiphospholipid antibody-induced fetal loss. J Exp Med. 2002 Jan 21;195(2):211-20. doi: 10.1084/jem.200116116. PMID 11805148
- [Background] Lockshin MD, Kim M, Laskin CA, Guerra M, Branch DW, Merrill J, Petri M, Porter TF, Sammaritano L, Stephenson MD, Buyon J, Salmon JE. Prediction of adverse pregnancy outcome by the presence of lupus anticoagulant, but not anticardiolipin antibody, in patients with antiphospholipid antibodies. Arthritis Rheum. 2012 Jul;64(7):2311-8. doi: 10.1002/art.34402. PMID 22275304
- [Background] Buyon JP, Kim MY, Guerra MM, Laskin CA, Petri M, Lockshin MD, Sammaritano L, Branch DW, Porter TF, Sawitzke A, Merrill JT, Stephenson MD, Cohn E, Garabet L, Salmon JE. Predictors of Pregnancy Outcomes in Patients With Lupus: A Cohort Study. Ann Intern Med. 2015 Aug 4;163(3):153-63. doi: 10.7326/M14-2235. PMID 26098843
- [Background] Kim MY, Buyon JP, Guerra MM, Rana S, Zhang D, Laskin CA, Petri M, Lockshin MD, Sammaritano LR, Branch DW, Porter TF, Merrill JT, Stephenson MD, Gao Q, Karumanchi SA, Salmon JE. Angiogenic factor imbalance early in pregnancy predicts adverse outcomes in patients with lupus and antiphospholipid antibodies: results of the PROMISSE study. Am J Obstet Gynecol. 2016 Jan;214(1):108.e1-108.e14. doi: 10.1016/j.ajog.2015.09.066. Epub 2015 Sep 29. PMID 26432463
- [Background] Yelnik CM, Laskin CA, Porter TF, Branch DW, Buyon JP, Guerra MM, Lockshin MD, Petri M, Merrill JT, Sammaritano LR, Kim MY, Salmon JE. Lupus anticoagulant is the main predictor of adverse pregnancy outcomes in aPL-positive patients: validation of PROMISSE study results. Lupus Sci Med. 2016 Jan 12;3(1):e000131. doi: 10.1136/lupus-2015-000131. eCollection 2016. PMID 26835148
- [Background] Yelnik CM, Porter TF, Branch DW, Laskin CA, Merrill JT, Guerra MM, Lockshin MD, Buyon JP, Petri M, Sammaritano LR, Stephenson MD, Kim MY, Salmon JE. Brief Report: Changes in Antiphospholipid Antibody Titers During Pregnancy: Effects on Pregnancy Outcomes. Arthritis Rheumatol. 2016 Aug;68(8):1964-9. doi: 10.1002/art.39668. PMID 26990620
- [Background] Buyon JP, Kim MY, Guerra MM, Lu S, Reeves E, Petri M, Laskin CA, Lockshin MD, Sammaritano LR, Branch DW, Porter TF, Sawitzke A, Merrill JT, Stephenson MD, Cohn E, Salmon JE. Kidney Outcomes and Risk Factors for Nephritis (Flare/De Novo) in a Multiethnic Cohort of Pregnant Patients with Lupus. Clin J Am Soc Nephrol. 2017 Jun 7;12(6):940-946. doi: 10.2215/CJN.11431116. Epub 2017 Apr 11. PMID 28400421
- [Background] Kim MY, Guerra MM, Kaplowitz E, Laskin CA, Petri M, Branch DW, Lockshin MD, Sammaritano LR, Merrill JT, Porter TF, Sawitzke A, Lynch AM, Buyon JP, Salmon JE. Complement activation predicts adverse pregnancy outcome in patients with systemic lupus erythematosus and/or antiphospholipid antibodies. Ann Rheum Dis. 2018 Apr;77(4):549-555. doi: 10.1136/annrheumdis-2017-212224. Epub 2018 Jan 25. PMID 29371202
- [Background] Hong S, Banchereau R, Maslow BL, Guerra MM, Cardenas J, Baisch J, Branch DW, Porter TF, Sawitzke A, Laskin CA, Buyon JP, Merrill J, Sammaritano LR, Petri M, Gatewood E, Cepika AM, Ohouo M, Obermoser G, Anguiano E, Kim TW, Nulsen J, Nehar-Belaid D, Blankenship D, Turner J, Banchereau J, Salmon JE, Pascual V. Longitudinal profiling of human blood transcriptome in healthy and lupus pregnancy. J Exp Med. 2019 May 6;216(5):1154-1169. doi: 10.1084/jem.20190185. Epub 2019 Apr 8. PMID 30962246
- [Background] Kaplowitz ET, Ferguson S, Guerra M, Laskin CA, Buyon JP, Petri M, Lockshin MD, Sammaritano LR, Branch DW, Merrill JT, Katz P, Salmon JE. Contribution of Socioeconomic Status to Racial/Ethnic Disparities in Adverse Pregnancy Outcomes Among Women With Systemic Lupus Erythematosus. Arthritis Care Res (Hoboken). 2018 Feb;70(2):230-235. doi: 10.1002/acr.23263. Epub 2017 Dec 29. PMID 28480528
- [Derived] Davis-Porada J, Kim MY, Guerra MM, Laskin CA, Petri M, Lockshin MD, Sammaritano LR, Branch DW, Sawitzke A, Merrill JT, Buyon JP, Salmon JE. Low frequency of flares during pregnancy and post-partum in stable lupus patients. Arthritis Res Ther. 2020 Mar 19;22(1):52. doi: 10.1186/s13075-020-2139-9. PMID 32188491
- [Derived] Yelnik CM, Lambert M, Drumez E, Le Guern V, Bacri JL, Guerra MM, Laskin CA, Branch DW, Sammaritano LR, Morel N, Guettrot-Imbert G, Launay D, Hachulla E, Hatron PY, Salmon JE, Costedoat-Chalumeau N. Bleeding complications and antithrombotic treatment in 264 pregnancies in antiphospholipid syndrome. Lupus. 2018 Sep;27(10):1679-1686. doi: 10.1177/0961203318787032. Epub 2018 Jul 17. PMID 30016929
- [Derived] Andrade D, Kim M, Blanco LP, Karumanchi SA, Koo GC, Redecha P, Kirou K, Alvarez AM, Mulla MJ, Crow MK, Abrahams VM, Kaplan MJ, Salmon JE. Interferon-alpha and angiogenic dysregulation in pregnant lupus patients who develop preeclampsia. Arthritis Rheumatol. 2015 Apr;67(4):977-87. doi: 10.1002/art.39029. PMID 25603823
- [Derived] Michael D Lockshin, Cohn E, Aslam A, Buyon JP, Salmon JE. Sex ratios among children of lupus pregnancies. Arthritis Rheum. 2013 Jan;65(1):282. doi: 10.1002/art.37718. No abstract available. PMID 23044629
- [Derived] Salmon JE, Heuser C, Triebwasser M, Liszewski MK, Kavanagh D, Roumenina L, Branch DW, Goodship T, Fremeaux-Bacchi V, Atkinson JP. Mutations in complement regulatory proteins predispose to preeclampsia: a genetic analysis of the PROMISSE cohort. PLoS Med. 2011 Mar;8(3):e1001013. doi: 10.1371/journal.pmed.1001013. Epub 2011 Mar 22. PMID 21445332
- See also: Clinical Trials at Hospital for Special Surgery — http://www.hss.edu/clinical-trials.asp
- See also: The PROMISSE Study: The Nation's Largest Ever Investigation of Pregnancy Loss in Lupus — http://www.hss.edu/conditions_promisse-largest-investigation-lupus-pregnancy-loss.asp
- See also: Pregnancy Safe for 80% of Women with Lupus — http://www.disabled-world.com/health/autoimmunediseases/lupus/pregnancy-hope.php
- See also: PROMISSE: progress in understanding pregnancy complications in patients with SLE — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3467516/
- See also: Lupus Anticoagulant Affects Pregnancy Outcomes — http://www.lupus.org/research-news/entry/lupus-anticoagulant-affects-pregnancy-outcomes